CLINICAL TRIAL: NCT06438874
Title: Type 2 Diabetes Post Exercise Arterial Stiffness
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss of funding.
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY2024-0610
Record Dates: First submitted 2024-05-23; First posted 2024-06-03 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exercise Test

STUDY DESIGN:
Intervention Model Description: The study will involve individuals diagnosed with type 2 diabetes mellitus (T2DM) who are currently receiving treatment with a glucagon-like peptide 1 (GLP1) agonist compared to a control group of individuals diagnosed with type 2 diabetes mellitus (T2DM) who are receiving treatment with drugs other than glucagon-like peptide 1 (GLP1) agonists. The study will not involve changes to medications for the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GLP-1 Treatment (Experimental): Individuals diagnosed with type 2 diabetes mellitus (T2DM) who are currently receiving treatment with a glucagon-like peptide 1 (GLP1) agonist.
  Interventions: Other: Exercise Test

INTERVENTIONS:
Other: Exercise Test — Exercise capacity will be measured as peak oxygen consumption (peakVO2) using an incremental exercise test on a cycle ergometer with an open-circuit spirometry system (TrueOne, Parvo Medics, Sandy, UT) to analyze expired gases. Exercise testing will follow the American College of Sports Medicine and American Heart Association guidelines. The investigators will use a graded protocol, starting with a warm-up at 0 watts for 5 minutes, followed by 15 watt increments every 2 minutes until volitional fatigue.

SUMMARY:
The overall aim of this research proposal is to determine the impact of GLP1 agonists on post-exercise arterial stiffness. Therefore, the investigators will examine the cardiovascular responses to exercise in individuals with Type 2 Diabetes mellitus (T2DM) taking these medications during and following a graded maximal exercise test.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is a significant public health concern associated with increased cardiovascular morbidity and mortality. Notably, individuals with T2DM often exhibit increased arterial stiffness, a key indicator of cardiovascular risk. Pharmacological interventions such as GLP1 agonists have emerged as crucial treatments for T2DM, offering glycemic control and potential cardiovascular benefits, including improvements in blood pressure and arterial stiffness. However, while the effects of GLP1 agonists on glycemic control and blood pressure regulation have been explored, their impact on arterial stiffness, specifically in response to exercise, remains largely unexplored in individuals with T2DM. Arterial stiffness is a critical marker of cardiovascular health, and its reduction is associated with decreased cardiovascular risk which include lowered blood pressure. Therefore, the overall aim of this research is to investigate whether GLP1 agonists attenuate arterial stiffness post exercise and reduce peak exercise blood pressure in individuals with T2DM.

ELIGIBILITY:
Inclusion Criteria:

Individuals diagnosed with type 2 diabetes mellitus (T2DM).

* Age between 18 and 60 years old.
* Currently receiving treatment with a glucagon-like peptide 1 (GLP1) agonist for the management of T2DM for a minimum duration of six months.
* For control group no current use of a glucagon-like peptide 1 (GLP1) agonist for the management of type 2 diabetes mellitus (T2DM).
* HbA1c levels between 6.5-8%
* Body Mass Index (BMI) within the range of 25 to 40 kg/m2.

Exclusion Criteria:

* Coronary heart disease.
* Pulmonary disease (e.g. asthma, chronic obstructive pulmonary disease)
* Neurological disorders (e.g. Alzheimer's disease, dementia)
* Congestive heart failure.
* Peripheral vascular disease.
* Liver failure.
* Kidney failure.
* Alcohol abuse.
* Drug abuse.
* Smoking.
* Hypertension (defined as Systolic Blood Pressure ≥ 140 mmHg or Diastolic Blood Pressure ≥ 90 mmHg)
* Insulin therapy for the management of T2DM
* Severe obesity (defined as Body Mass Index >40 kg/m2);
* Pregnancy
* Non-English speaking individuals

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Arterial stiffness | Baseline and up to 20 minutes post exercise
  Measured via pulse wave velocity

SECONDARY OUTCOMES:
Blood pressure | Through exercise test completion, an average of 10 minutes
  Peak exercise blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Ronald E Jackson, PhD, Principal Investigator — University of Illinois Chicago

IPD SHARING:
Plan to Share IPD: No